CLINICAL TRIAL: NCT07123701
Title: A Randomized Placebo-controlled Clinical Trial of Tanshinone Capsules in the Treatment of Patients With COVID-19
Brief Title: Clinical Study of Tanshinone Capsules Against COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Liu Shuwen (Other)
Responsible Party: Sponsor-Investigator, Liu Shuwen, professor, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Southern MUC
Record Dates: First submitted 2025-08-11; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
MeSH Terms: conditions — COVID-19 | interventions — tanshinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- placebo-controlled clinical trial of tanshinone capsules in the treatment of patients with COVID-19 (Experimental): The experimental group was given tanshinone capsule, and the placebo control was given tanshinone capsule placebo, orally administered 3 times a day, 4 capsules/time, 0.25g/ capsule, for 5 days.
  Interventions: Drug: Tanshinone capsules

INTERVENTIONS:
Drug: Tanshinone capsules — Tanshinone capsules were used in this intervention for COVID-19 patients

SUMMARY:
The variation of SARS-CoV-2 has caused many countries to face the problem of multiple outbreaks. Gene mutations can change the transmicity, pathogenicity, and immunogenicity of the virus. For example, the Omicron variant circulating around the world spreads faster, increases infectivity, and infects a younger population, which in turn affects the efficacy of antiviral drugs or weakens the protective efficiency of vaccines. Therefore, in order to fully respond to the variation of SARS-CoV-2 and possible new coronaviruses in the future, the development of broad-spectrum anti-coronavirus drugs is an urgent clinical need. Tanshinone capsule is a marketed drug, which is made of the lipid-soluble components of the root of Danshen, a traditional Chinese medicine. It is used for anti-bacterial and anti-inflammatory functions, and is used for acne, tonsillitis and furunils. Its clinical use relives the situation of antibiotic resistance and toxicity. Our previous basic research has shown that tanshinone capsules have anti-SARS-CoV-2 activity in vitro and in humanized ACE2 transgenic mice. The use of tanshinone capsules in the treatment of SARS-CoV-2 infection can further broaden the antiviral pharmacological activity of tanshinone capsules and may increase its clinical function as an antiviral drug for the treatment of viral infection. On the one hand, tanshinone capsules are oral traditional Chinese medicine capsules, which have the advantages of low production/transportation cost, high safety and high patient compliance. On the other hand, tanshinone capsules are expected to reduce the level of inflammation in patients and improve the symptoms of COVID-19 while preventing and treating COVID-19 infection. It can meet the major needs of novel coronavirus pneumonia drug research and development to a high degree.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnosis of SARS-CoV-2 infection issued by the National Health Commission of the People's Republic of China (Trial Version 10). Based on the etiology or serological test, within 2 days of diagnosis, and meet the following conditions: 1) The Ct values of N gene and ORF gene of 2019-ncov infection were both less than 30 (fluorescence quantitative PCR method, the cut-off value was 40); 2) Mild and/or moderate clinical classification: subjects had at least one or more of the following clinical symptoms of COVID-19 with a symptom score ≥1 at the time of screening, including but not limited to: fever, cough, sore throat, nasal congestion or runny nose, headache, muscle pain, nausea, vomiting, diarrhea, shortness of breath or dyspnea, chills or chills.
2. Age of 18-65 years old, both sexes;
3. Participants were required to meet one or more of the following criteria: 1) ≤3 days from the first administration of the investigational drug to the positive SARS-CoV-2 virus infection test specimen during the screening period, 2) ≤3 days from the first onset of COVID-19 symptoms to the first administration of the investigational drug;
4. Patients voluntarily participated in this study, and they or their legal representatives signed written informed consent and were willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients at high risk of severe or critical illness and diagnosed as severe or critical illness before entering the study according to the "Diagnosis and Treatment Protocol for novel coronavirus Infection (Trial version 10)";
2. Received antiviral treatment before study entry, such as Chinese patent medicine or Chinese medicine formula treatment, Paxlovid, ritonavir tablets, SARS-CoV-2 monoclonal antibody treatment, convalescent plasma of convalescent patients, other clinical trial drugs indicated for COVID-19, etc. (except previous treatment for COVID-19 infection);
3. Subjects with known allergy to therapeutic drug tanshinone capsules or allergic constitution (including susceptible to allergic reactions to other drugs);
4. Suffering from diseases that seriously affect the immune system, such as human immunodeficiency virus (HIV) infection, or blood system, or splenectomy, organ transplantation, etc.
5. Pregnant and lactating women;
6. Suspected bacterial, fungal, viral or other infections other than SARS-CoV-2 during the screening period;
7. Patients with bronchopneumonia, chronic lung abscess, chronic cough for more than 8 weeks, chronic pharyngitis with cough and other diseases before entering the study;
8. One of the following conditions during the screening period: 1) ALT or AST>1.5 times ULN; 2) eGFR<60mL/min; 3) hemoglobin <8.0g/L, platelet <5000/μL;
9. Patients who participated in other clinical trials within the past 3 months;
10. Persons not eligible for enrollment at the investigator's discretion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Negative conversion time of nucleic acid in throat swab | After the screening period, the first day of dosing was day 1
  The task turned negative when the CT value of ORF1ab gene and N gene was greater than 30

CONTACTS AND LOCATIONS:
Overall Officials: guodong G HU, DOCTOR, Principal Investigator — Dongguan People's Hospital
Locations (1):
- Dongguan People's Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Gender, age, and bmi
Supporting Information: ICF
Time Frame: 2025.8.1-2028.1.1
Access Criteria: ifc

DOCUMENTS (2):
  • Study Protocol (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT07123701/Prot_000.pdf
  • Informed Consent Form (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT07123701/ICF_001.pdf